CLINICAL TRIAL: NCT03533478
Title: Efficacy of Nutritional Supplements Alzer® and Diamel® to Prevent Severe Diabetes Macular Edema. Clinical Trial Phase II.
Brief Title: Alzer® and Diamel® to Prevent Severe Diabetes Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALZER-DIAMEL-EMD-2014
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Macular Edema
Keywords: Nutritional supplement; Diabetic Macular Edema; Diabetes; Alzer; Oxidative Stress; Diamel
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): 32 patients with mild or moderate diabetic macular edema.
  Interventions: Dietary Supplement: Oral treatment Alzer y Diamel
- Group II (Placebo Comparator): 32 patients with mild or moderate diabetic macular edema
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral treatment Alzer y Diamel — Alzer:
  Administration way: Oral Dosage: one 500 mg tablet 3 times a day (1500 mg daily) Frequency: after breakfast, lunch and dinner. Duration: one year.
  Diamel:
  Administration way: Oral Dosage: two 660mg capsules 3 times a day (3960 mg daily) Frequency: before breakfast, lunch and dinner. Duration: one year.
  Arms: Group I
Dietary Supplement: Placebo — Placebo treatment
  Arms: Group II

SUMMARY:
Macular edema is the main cause of low vision in diabetics. They continue looking for new treatment alternatives. The nutritional supplement Alzer, is a powerful antioxidant that together with Diamel, a supplement that has shown efficacy in metabolic control, could be a therapeutic option. Objective: To evaluate the therapeutic efficacy of the Alzer Diamel combination in mild and moderate macular edema. Material and method: A randomized double-blind phase II clinical trial versus placebo will be conducted in 64 patients, who will be randomly assigned to two groups, one will receive Alzer + Diamel and another will receive placebo from Alzer and Diamel. All patients will undergo clinical, biochemical and ophthalmological evaluation during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics type 2 insulin treated.
* Age between 18 and 65 years.
* Glycosylated hemoglobin (HB A1c) <8% at the beginning of the investigation.
* Patients who express written voluntariness to enter the study with their signature of the informed consent document.
* If woman of childbearing age, negative pregnancy test and use of barrier contraceptives.

Exclusion Criteria:

* Pregnancy and lactation.
* Age over 65 years.
* Macular edema with vitreous-retinal traction or other cause (renal, arterial hypertension, post-surgical).
* Opacity of the refractive media that hinders the ophthalmological examination.
* History of hypersensitivity to another similar product or one of its components.
* Patients at potential risk of not compliance the study (those who will travel during the period of the investigation or distance in their residence, outside the city).
* Subjects who are participating in another clinical trial Patients with cognitive disorders or a mental disorder that hinders their follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Macular retinal thickness | 1 year
  macular retinal measure

SECONDARY OUTCOMES:
Visual acuity | 1 year
  visual acuity test

CONTACTS AND LOCATIONS:
Overall Officials: Juana Elvira Maciques Rodríguez, Dr., Principal Investigator — National Institute of Endocrinology, Cuba
Locations (1):
- National Institute of Endocrinology, Vedado, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code